CLINICAL TRIAL: NCT00745251
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study of VI-0521 for the Treatment of Obstructive Sleep Apnea / Hypopnea Syndrome in Obese Adults
Brief Title: A Study of VI-0521 for the Treatment of Obstructive Sleep Apnea / Hypopnea Syndrome in Obese Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OB-204
Record Dates: First submitted 2008-08-31; First posted 2008-09-03 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-09

CONDITIONS: Sleep Apnea
Keywords: Sleep apnea; obesity
MeSH Terms: conditions — Sleep Apnea Syndromes; Obesity | interventions — Qnexa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VI-0521 (Experimental): 15 mg Phentermine and 92 mg Topiramate
  Interventions: Drug: VI-0521
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: VI-0521 — 15 mg Phentermine and 92 mg Topiramate
  Other Names: Qnexa; PHEN/TPM
  Arms: VI-0521
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to evaluate the safety and efficacy of VI-0521 compared to placebo in the treatment of obese adults with obstructive sleep apnea (OSA) and to assess the relative contributions of weight loss on parameters of OSA in these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Obese adults 30 - 65 years old (inclusive);
* Women of child-bearing potential must be using adequate contraception;
* BMI between 30 and 40 kg/m2 (inclusive);
* Diagnosis of OSA syndrome with Apnea/Hypopnea Index (AHI) of 15 or greater;
* Unwilling or unable to comply with CPAP treatment;

Exclusion Criteria:

* Known allergy or hypersensitivity to phentermine or topiramate;
* Sleep disorder other than OSA syndrome;
* Women who are pregnant, breast feeding, or intend to become pregnant during the study;
* Presence of unstable angina or heart failure corresponding to NYHA functional class III or IV;
* History of myocardial infarction or coronary revascularization within the past year; any history of stroke;
* Presence of any clinically significant abnormality on electrocardiogram;
* Use of any prescription CNS stimulants;
* History of cholecystitis or cholelithiasis unless treated by cholecystectomy;
* History of glaucoma or any past or present use of medications to treat increased intraocular pressure;
* Weight gain or loss of greater than 5 kg, use of a very low-calorie diet, or participation in a formal weight loss program (investigational or otherwise) within the past 3 months;
* Previous bariatric surgery;
* Shift workers or any subjects with a circadian rhythm disorder;
* Professional drivers or commercial pilots;
* History of nephrolithiasis;
* More than one lifetime episode of major depression;
* History of bipolar disorder, obsessive compulsive disorder, borderline personality disorder, psychotic depression, schizophrenia, schizoaffective disorder, or any other psychotic disorder; history of any psychiatric hospitalization;
* History of a seizure disorder; concurrent use of any anticonvulsant drug (other than assigned study drug);

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bowden, MD, Study Director — VIVUS LLC
Locations (1):
- Kentucky Research Group, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred in 1 investigative site in the U.S. between August 2008 to February 2009
Groups:
- Top Dose: PHEN/TPM 15mg/92mg
Period: Overall Study
Arm/Group | Placebo | Top Dose
Started | 23 | 22
Completed | 21 | 19
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Top Dose | Total
Number analyzed (Participants) | 23 | 22 | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 51.4 (5.74) | 53.4 (6.95) | 52.4 (6.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 15 | 9 | 24
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in the Apnea/Hypopnea Index (AHI) Between Baseline and Week 28/Early Term.
Description: AHI is calculated as the mean number of apnea or hypopnea episodes (each lasting a minimum of 10 second) observed per hour of sleep
Time Frame: between baseline and Week 28
Population: Intent-to-treat Last-observation-carried-forward (ITT-LOCF)
Measure: Least Squares Mean (Standard Error); unit: events/hour
Arm/Group | Placebo | Top Dose
Number analyzed (Participants) | 23 | 22
events/hour | -16.6 (4.15) | -31.46 (4.25)
Statistical Analysis 1: Comparison: Placebo vs Top Dose; Test type: Superiority or Other; p = 0.0084, ANCOVA; Mean Difference (Final Values) = -14.86, 95% CI 1-sided [upper limit -4.84], Standard Error of Mean 5.95

2. Secondary Outcome: Percent Change in Weight From Baseline to Week 28
Time Frame: baseline to week 28
Population: Intent-to-treat Last-observation-carried-forward (ITT-LOCF)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Top Dose
Number analyzed (Participants) | 23 | 22
percent change | -10.26 (1.17) | -4.21 (1.15)
Statistical Analysis 1: Comparison: Placebo vs Top Dose; Test type: Superiority or Other; p = 0.0006, ANCOVA; Mean Difference (Final Values) = -6.05, 95% CI 2-sided [-9.37 to -2.74], Standard Error of Mean 1.64

ADVERSE EVENTS:
Time Frame: AEs were collected from when written informed consent was provided through 28 days after the last dose of investigational product.
Arm/Group | Placebo | Top Dose
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/22
Other Adverse Events (participants affected / at risk) | 17/23 | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | Top Dose (N=22)
cerebrovascular accident (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | Top Dose (N=22)
tinnitus (Ear and labyrinth disorders) | 0 | 2
constipation (Gastrointestinal disorders) | 2 | 3
diarrhea (Gastrointestinal disorders) | 2 | 3
dry mouth (Gastrointestinal disorders) | 0 | 11
nausea (Gastrointestinal disorders) | 1 | 2
disturbance in attention (Nervous system disorders) | 1 | 2
dysgeusia (Nervous system disorders) | 0 | 6
headache (Nervous system disorders) | 0 | 2
hypoaesthesia (Nervous system disorders) | 0 | 3
parethesia (Nervous system disorders) | 0 | 3
somnolence (Nervous system disorders) | 2 | 1
feeling jittery (General disorders) | 0 | 2
keratitis (Eye disorders) | 0 | 1
vision blurred (Eye disorders) | 0 | 1
gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
gingival bleeding (Gastrointestinal disorders) | 0 | 1
gingival pain (Gastrointestinal disorders) | 0 | 1
hematochezia (Gastrointestinal disorders) | 0 | 1
hemorrhoids (Gastrointestinal disorders) | 0 | 1
chest discomfort (General disorders) | 0 | 1
irritability (General disorders) | 1 | 1
mucosal dryness (General disorders) | 0 | 1
gastroenteritis viral (Infections and infestations) | 4 | 2
nasopharyngitis (Infections and infestations) | 1 | 3
sinusitis (Infections and infestations) | 0 | 5
tonsillitis (Infections and infestations) | 0 | 1
upper respiratory tract infection (Infections and infestations) | 1 | 4
viral upper respiratory tract infection (Infections and infestations) | 0 | 1
hand fracture (Injury, poisoning and procedural complications) | 0 | 1
procedural pain (Injury, poisoning and procedural complications) | 0 | 1
food craving (Metabolism and nutrition disorders) | 1 | 1
back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
amnesia (Nervous system disorders) | 0 | 1
dizziness (Nervous system disorders) | 0 | 1
parosmia (Nervous system disorders) | 0 | 1
tremor (Nervous system disorders) | 0 | 1
agitation (Psychiatric disorders) | 0 | 1
mood altered (Psychiatric disorders) | 0 | 1
sleep disorder (Psychiatric disorders) | 0 | 1
stress (Psychiatric disorders) | 0 | 1
dysuria (Renal and urinary disorders) | 0 | 1
nephrolithiasis (Renal and urinary disorders) | 0 | 1
nocturia (Renal and urinary disorders) | 0 | 1
urinary hesitation (Renal and urinary disorders) | 0 | 1
perineal cyst (Reproductive system and breast disorders) | 0 | 1
allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
rash (Skin and subcutaneous tissue disorders) | 0 | 1
flushing (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's written notification that publication of results is no longer planned or 12 months after termination of the study at all sites, Institution & PI may publish, upon written approval from Sponsor, results of the Study. Sponsor will be given the opportunity to review any proposed publication at least 60 days prior to submission for publication or disclosure. Upon Sponsor's written request, Institution and PI shall not publish or disclose information related to the Study.